CLINICAL TRIAL: NCT02145637
Title: Phase I Study of the Combination of Afatinib and Ruxolitinib in Patients With Treatment-refractory Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0405
Record Dates: First submitted 2014-04-23; First posted 2014-05-23 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2018-03

CONDITIONS: NSCLC
Keywords: Cancer, Lung cancer, Head and neck squamous cell carcinoma, Afatinib, Ruxolitinib, EGFR, JAK, STAT
MeSH Terms: conditions — Neoplasms; Lung Neoplasms | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Afatinib plus Ruxolitinib combination (single arm) (Experimental)
  Interventions: Drug: Afatinib plus Ruxolitinib combination therapy

INTERVENTIONS:
Drug: Afatinib plus Ruxolitinib combination therapy

SUMMARY:
This phase Ib study will investigate dose limiting toxicity (DLT) and maximum tolerated dose (MTD) of afatinib and ruxolitinib combination therapy, based on the preclinical data that inhibition of IL-6R/JAK1 signal transmission pathway will increase sensitivity to afatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Stage 4 NSCLC patients
2. disease progression after platinum doublet (all), EGFR TKI (if EGFR mutant), and crizotinib (if ALK positive)
3. Men and women aged 20 years or older
4. Recovery from previous drug-related toxicity: CTCAE 4.03 ≤ Grade 1
5. ECOG 0 or 1
6. able to orally take and retain drug
7. have a measurable or unmeasurable lesion under RECIST 1.1 Criteria
8. have proper hematological, renal, and hepatic functions
9. intention to use an acceptable contraception
10. able to read and understand the informed consent form

Exclusion Criteria:

1. previous chemotherapy, radiation therapy, immunotherapy, or other anticancer therapy within 14 days
2. Clinically significant gastrointestinal disorder or malabsorption syndrome
3. Acute digestive disorder
4. major organ failure
5. Significant cardiac disorders
6. major operation of a main organ in 4 weeks
7. Untreated symptomatic brain metastasis
8. pregnant or nursing
9. previously diagnosed Interstitial lung disease(ILD)
10. previously treated with irreversible pan-HER inhibitor including Afatinib or Ruxolitinib
11. previously experienced hypersensitivity to an ingredient of the study drug
12. must receive CYP3A4 inducer or inhibitor persistently during the study period.
13. HIV positive or active hepatitis
14. threatening patient's safety is predicted

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05-07; Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
To set a recommended phase II dose (RP2D) | 36 days
  We will set a recommended phase II dose (RP2D) using conventional 3+3 deisgn.

SECONDARY OUTCOMES:
Safety and tolerability (dose relating toxicity; DLT) | 1year
  Adverse events (AEs) will be assessed according to NCI common toxicity criteria (CTC) version 4.03.
Overall response rate (ORR) | 1year
  Response and progression will be evaluated in this study using modified international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
Progression free survival (PFS) | 1year
  PFS will be defined as the start of the treatment to the first occurrence of progression, relapse, or death from any cause as assessed by the investigator.
Overall survival (OS) | 1year
  OS will be defined as the start of the treatment to the date of death due to any cause.
Pharmacodynamic biomarker | 1year
  The biomarkers marker related with EGFR and JAK/STAT pathway as well as gene analysis, using peripheral blood mononuclear cell(PBMC), circulating tumor cell (CTC) and skin and tumor tissue sample will be analyzed.

REFERENCES:
- [Derived] Park JS, Hong MH, Chun YJ, Kim HR, Cho BC. A phase Ib study of the combination of afatinib and ruxolitinib in EGFR mutant NSCLC with progression on EGFR-TKIs. Lung Cancer. 2019 Aug;134:46-51. doi: 10.1016/j.lungcan.2019.05.030. Epub 2019 May 28. PMID 31319994